CLINICAL TRIAL: NCT04764656
Title: Observational Study to Evaluate Fluid Resolution and Effectiveness of Brolucizumab for Neovascular Age-related Macular Degeneration (nAMD) in Portugal
Brief Title: Observational Study to Evaluate Fluid Resolution and Effectiveness of Brolucizumab for nAMD in Portugal
Acronym: BLUESKY-PT
Status: Terminated | Type: Observational
Why Stopped: The study was terminated earlier since the obtained sample was not representative of the Portuguese population, and pointed to the high fragility in evaluating the data, making it difficult to carry out a statistical study and draw valid conclusions.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CRTH258APT02
Record Dates: First submitted 2021-02-19; First posted 2021-02-21 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Neovascular Age-related Macular Degeneration (nAMD)
Keywords: Beovu; Brolucizumab; nAMD; non-interventional trial; fluid resolution
MeSH Terms: interventions — brolucizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Brolucizumab: Naïve (Patients being the first time treated) and pre-treated patients
  Interventions: Drug: Brolucizumab

INTERVENTIONS:
Drug: Brolucizumab — There is no treatment allocation. Patients administered Brolucizumab by prescription that have started before inclusion of the patient into the study will be enrolled.

SUMMARY:
This study is a prospective, observational, non-interventional, multicenter, open-label, single arm study in patients being treated for nAMD with brolucizumab in Portugal.

DETAILED DESCRIPTION:
Naïve and pre-treated patients will be included after decision to start treatment with brolucizumab and consent is given.

The baseline visit will be used to assess eligibility and collect baseline characteristics information. The study eye will be defined as the first eye treated during the study; the other eye will be considered as fellow eye. If both eyes are treated at baseline, the eye with the worse visual acuity will be chosen as the study eye (if the visual acuity is measured equal, the treating ophthalmologist defines the study eye upon his discretion). The follow-up visits will take place at a frequency defined as per investigator's discretion. Patients that have not received an intravitreal anti-VEGF injection or visited an eye specialist for at least 6 months will be discontinued from the observation.

Retrospective data will be collected for switch patients starting treatment with brolucizumab for up to six months before baseline. Patients, already being treated with brolucizumab may also be included. Here, retrospective data will be collected since the first brolucizumab injection.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of nAMD
2. Male and Female patients with ≥40 years of age at index
3. Receipt of at least one injection of brolucizumab during the recruitment period
4. Signed written informed consent

Exclusion Criteria:

1. Patients treated for RVO, DME, mCNV, and have diagnoses of diabetes-related macular degeneration within 6 months prior to the index date
2. Receipt of any anti-VEGF treatment other than brolucizumab in the study eye at index date
3. Central subfield of the study eye affected by fibrosis or geographic atrophy or total area of fibrosis >50% of the total lesion in the study eye at Screening
4. Any active intraocular or periocular infection or active intraocular inflammation in either eye at index date
5. Patients who have been on anti-VEGF treatment for longer than 3 years (before index date)
6. Patients that have any contraindication and are not eligible for treatment with brolucizumab as according to the SmPC
7. Any medical or psychological condition in the treating physician's opinion which may prevent the patient from the 24 months study participation
8. Patients participating in parallel in an interventional clinical trial
9. Patients participating in parallel in any other NIS generating primary data for an anti-VEGF drug
10. Retinal pigment epithelial rip/tear in the study eye at Screening or Baseline or current vitreous hemorrhage or history of vitreous hemorrhage in the study eye within 4 weeks prior to Baseline
11. Subretinal blood affecting the foveal center point and/or >50% of the lesion of the study eye at Screening

Ages: 40 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include an estimated number of 120 naïve patients and 180 switch patients with a diagnosis of nAMD being treated with brolucizumab in private clinics in Portugal during the recruitment period
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-02-16 (Actual)

PRIMARY OUTCOMES:
Percentage of patients that are absent of subretinal fluid (SRF) and intra-retinal fluid (IRF) in the study eye | month 12
  This primary study objective will be addressed considering treatment naïve and pre-treated patient eyes included in the study, analyzed as two independent groups (naïve and switch).

SECONDARY OUTCOMES:
Fluid resolution after initiation of brolucizumab | month 24
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Visual Actuity (VA) change from baseline | Baseline, month 24
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Characterize Choroidal Neovascularization (CNV) morphology (BIRL) and activity | month 24
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Number of injections and total number of visits | month 24
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Describe the distribution of injection intervals | month 24
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Number of Spectral Contrast Optical Coherence Tomography (SC-OCTs) done | month 24
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Characterize the patients switching to another antivascular endothelial growth factor (anti-VEGF) | month 24
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Discontinuation rate | month 24
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Assess the safety of brolucizumab | month 24
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- Portugal (6):
  - Novartis Investigative Site, Funchal
  - Novartis Investigative Site, Leiria
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
  - Novartis Investigative Site, Santa Maria da Feira
  - Novartis Investigative Site, Tomar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CRTH258APT02 from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18270